CLINICAL TRIAL: NCT04109131
Title: A Brain Metastases Research Platform to Tackle the Challenge of CNS Metastases in Solid Tumours - BrainStorm Program
Brief Title: A Brain Metastases Research Platform to Tackle the Challenge of CNS Metastases in Solid Tumours
Acronym: BrainStorm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Fondation Cancer, Belgique (Unknown); Les Amis (Unknown); Bristol-Myers Squibb (Industry); Fondation Cancer, Luxembourg (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IJB-BS-ODN-006
Record Dates: First submitted 2019-07-12; First posted 2019-09-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: CNS Metastases
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNS metastases from solid tumours (Other): The study will be organised on three time-periods based on the time of the 1st CNS event:
  Part A - Pre-diagnosis period: before diagnosis of the 1st CNS event Part B - At 1st CNS diagnosis period Part C - Post diagnosis period: after the 1st CNS event
  Interventions: Other: Samples collection: Plasma; Other: Samples collection: CSF; Other: Samples collection: Non-CNS Metastatic Tumour Tissue; Other: Brain MRI; Other: Samples collection: Serum

INTERVENTIONS:
Other: Samples collection: Plasma — At baseline
  Part A:
  * TNBC/ HER2+ BC: once a year
  * NSCLC/SCLC: every 4 months
  * Melanoma: every 6 months
  Part B:
  o As close as possible to the diagnosis of CNS metastases and no later than 6 weeks after diagnosis
  Part C:
  o Every 3 months (+/- 1 month)
  Other Names: Blood for plasma preparation
Other: Samples collection: CSF — Part B: Mandatory CSF sampling at CNS diagnosis when clinically possible unless medically contra-indicated - As close as possible to the diagnosis of CNS metastases and no later than 6 weeks after diagnosis Part C: Additional CSF sampling in case CSF sampling is performed for routine clinical practice
  Other Names: CSF sample
Other: Samples collection: Non-CNS Metastatic Tumour Tissue — Part B: Highly recommended non-CNS metastatic tumour tissue collection (1FFPE and 1 FT) at CNS metastases diagnosis (Part B) (NB: Bone lesions are excluded) - As close as possible to the diagnosis of CNS metastases and no later than 6 weeks after diagnosis
  Other Names: Non-CNS Metastatic Tumour Tissue collection
Other: Brain MRI — Part A:
  * Brain MRI at inclusion is allowed within 45 days before enrolment
  * Brain MRI pre-CNS diagnosis (Part A) : HER2 BC/TNBC: once a year; NSCLC/SCLC: every 4 months; Melanoma: every 6 months (+/- 1 month)
  Part B:
  o As close as possible to the diagnosis of CNS metastases and no later than 6 weeks after diagnosis
  Part C:
  o Brain MRI post-CNS diagnosis (Part C): every 3 months (+/- 1 month window)
Other: Samples collection: Serum — At baseline
  Part A:
  * TNBC/ HER2+ BC: once a year
  * NSCLC/SCLC: every 4 months
  * Melanoma: every 6 months
  Part B:
  o As close as possible to the diagnosis of CNS metastases and no later than 6 weeks after diagnosis for cohorts 1-5.
  Other Names: Blood for serum preparation

SUMMARY:
Despite some encouraging data, systemic treatment of CNS metastases from solid tumors remains experimental.

Better knowledge on the evolving epidemiology and biology of BM are key elements for the development of new treatment strategies and identification of promising therapeutic targets for new compounds. Further biological findings may help to better understand the heterogeneity between the primary tumor and the CNS metastases and to identify new targets for therapy thus improving patients' outcome.

In this context, the Oncodistinct network and the Jules Bordet institute propose to build a multidisciplinary Brain Metastases Clinical Research Platform called BrainStorm. The BrainStorm program will focus on patients with newly diagnosed non-CNS metastatic solid tumors with high risk of developing CNS metastases and will allow building a large clinico pathological database for CNS metastases including ctDNA analyzes from CSF samples. Substudies will be proposed at each time-period with the final objective to develop innovative treatment approaches and strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
3. Female or Male
4. Eligible for part A: Subjects (from cohorts 1 to 5) with newly diagnosed or up to 24 months from diagnosis of non-CNS metastases. Enrolment of exceptional cases surpassing 24 months from diagnosis will be allowed for up to 20% of subjects enrolled with HER2+ BC (cohort 2) and NSCLC harbouring driver mutations (cohort 3).

   Eligible for part B: Subjects (from cohorts 1 to 7) presenting with a first CNS event and not yet enrolled in the program

   Seven cohorts of subjects are defined in this prospective multicenter study:
   * Cohort 1: Triple negative breast cancer (TNBC)
   * Cohort 2: HER 2 positive breast cancer (HER2+ BC)
   * Cohort 3: Non-small cell lung cancer (NSCLC)
   * Cohort 4: Small cell lung cancer (SCLC)
   * Cohort 5: Melanoma
   * Cohort 6: Other solid tumours (apart from the above mentioned subtypes
   * Cohort 7: Radiologically or cytologically confirmed leptomeningeal carcinomatosis
5. Availability of either primary and/or non-CNS metastatic archival tumour tissue is mandatory for inclusion.
6. Willingness to undergo lumbar puncture at diagnosis of CNS metastases unless medical contra-indications
7. Predicted life expectancy > 3 months.
8. Women of childbearing potential must have a negative urine pregnancy test done within 28 days prior to enrolment
9. Effective contraception is in place for women of childbearing potential
10. Completion of all necessary screening procedures within 28 days prior to enrolment.
11. Signed Informed Consent form (ICF) obtained prior to any study related procedure.

    Inclusion criterion applicable to FRANCE only
12. Affiliated to the French Social Security System

Exclusion Criteria:

1. Pregnant and/or lactating women.
2. Previous or current malignancies of other histologies within the last 2 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin.
3. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.

   Exclusion criterion applicable to FRANCE only
4. Vulnerable persons according to the article L.1121-6 of the Public Health Code, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Better understanding of the epidemiology of CNS metastases from solid tumours | through study completion, approximately 96 months
  To collect data regarding the epidemiology of CNS metastases from solid tumours and identify risk factors for CNS metastases development, including:
  * Time to the first CNS event
  * Time to the second CNS after first treatment and subsequent CNS events
Better understanding of the epidemiology of CNS metastases from solid tumours | through study completion, approximately 96 months
  To collect data regarding the epidemiology of CNS metastases from solid tumours and identify risk factors for CNS metastases development, including::
  - Time to whole brain radiotherapy
Better understanding of the epidemiology of CNS metastases from solid tumours | through study completion, approximately 96 months
  To collect data regarding the epidemiology of CNS metastases from solid tumours and identify risk factors for CNS metastases development, including:
  - Overall survival
Better understand the biology of CNS metastases (brain and leptomeningeal carcinomatosis) using CSF-ctDNA as a surrogate endpoint for CNS tumour tissue DNA. | through study completion, approximately 96 months
  To collect data regarding the biology of CNS metastases by investigating on:
  - Presence of CSF-ctDNA at diagnosis of CNS metastases
Better understand the biology of CNS metastases (brain and leptomeningeal carcinomatosis) using CSF-ctDNA as a surrogate endpoint for CNS tumour tissue DNA. | through study completion, approximately 96 months
  To collect data regarding the biology of CNS metastases by investigating on:
  - Presence of plasma ctDNA at diagnosis of CNS metastases
Better understand the biology of CNS metastases (brain and leptomeningeal carcinomatosis) using CSF-ctDNA as a surrogate endpoint for CNS tumour tissue DNA. | through study completion, approximately 96 months
  * quantification of plasma ctDNA and CSF-ctDNA using deep targeted NGS
  * deep targeted next-generation sequencing (NGS) on DNA samples from primary or non-CNS metastases as well as germline DNA samples and CNS metastases if surgery
Better understand the biology of CNS metastases (brain and leptomeningeal carcinomatosis) using CSF-ctDNA as a surrogate endpoint for CNS tumour tissue DNA. | through study completion, approximately 96 months
  - A set of 1-3 point mutations (single nucleotide variants) will be selected for each subject based on the above analyses for the identification and quantification of plasma ctDNA and CSF-ctDNA using deep targeted NGS
Better understand the biology of CNS metastases (brain and leptomeningeal carcinomatosis) using CSF-ctDNA as a surrogate endpoint for CNS tumour tissue DNA. | through study completion, approximately 96 months
  - Standard analyses cytology and biochemistry analyses
Better understand the biology of CNS metastases (brain and leptomeningeal carcinomatosis) using CSF-ctDNA as a surrogate endpoint for CNS tumour tissue DNA. | through study completion, approximately 96 months
  - Quantitative measurement of serum neuron-specific enolase

OTHER OUTCOMES:
Better understand the predictive value of NSE for the development of CNS metastases on subjects with newly diagnosed non-CNS metastatic solid tumours with high risk of developing CNS metastases. | through study completion, approximately 96 months
  To collect data regarding the biology of CNS metastases by investigating on :
  * Time to the first CNS event
  * Time to the second CNS event
  * Time to whole brain radiotherapy (WBR)
  * Time from the date of diagnosis of the first CNS event and the time of death by any cause
Better understand the predictive value of NSE for the development of CNS metastases on subjects with newly diagnosed non-CNS metastatic solid tumours with high risk of developing CNS metastases. | through study completion, approximately 96 months
  Levels of neuron specific enolase in blood
Better understand the predictive value of NSE for the development of CNS metastases on subjects with newly diagnosed non-CNS metastatic solid tumours with high risk of developing CNS metastases. | through study completion, approximately 96 months
  Deep targeted next-generation sequencing (NGS) on DNA samples from primary or non CNS metastases as well as germline DNA samples and CNS metastases if surgery. A set of 1-3 point mutations (single nucleotide variants) will be selected for each subject based on the above analyses for the identification and quantification of plasma ctDNA and CSF-ctDNA using deep targeted NGS. Subsequently targeted gene sequencing will be performed on DNA samples from CSF and plasma in case of at least 5% tumour mutant allele frequency (MAF) and CNS metastases in case of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Kotecki, MD, Study Chair — Jules Bordet Institute
Locations (17):
- Belgium (9):
  - Institut Jules Bordet, Anderlecht
  - Hôpital Erasme, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
  - CHU Ambroise Paré, Mons
  - CHU UCL Namur - Site de Sainte-Elisabeth, Namur
- France (7):
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - Institut Universitaire de Cancérologie AP-HP Sorbonne Université, Hopital Tenon, Paris
  - Institut Curie, Paris
  - Centre Henri Becquerel, Rouen
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer - Oncopole, Toulouse
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg